CLINICAL TRIAL: NCT07127601
Title: Comparative Study Between US Guided Erector Spinae and US Guided Cudal Epidural Block in Paediatric Unilateral Inguinal Hernia Repair Adjuvant to General Anaesthesia
Brief Title: Comparative Study Between US Guided Erector Spinae and US Guided Cudal Epidural Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Noser, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R 14 2022
Record Dates: First submitted 2024-06-14; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia; Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound guided erector spinae plain block (ESPB). (Experimental)
  Interventions: Procedure: Ultrasound guided erector spinae plain block (ESPB).
- caudal analgesia (anatomically)with lumber level of anagesia (Active Comparator)
  Interventions: Procedure: Ultrasound guided erector spinae plain block (ESPB).

INTERVENTIONS:
Procedure: Ultrasound guided erector spinae plain block (ESPB). — Depending on the size of patient, either a 27 g 3 cm hypodermic needle or a 21 g 5 or 10 cm short bevel needle was used. All blocks were performed with the ultrasound guidance in the parasagittal position and with continuous in-plane needle visualization. The local anesthetic was deposited in the fascial plane deep to the erector spinae muscle superficial to the transverse processes, after confirming the correct tissue plane by hydro-dissection. protocols for choosing 0.25% bupivacaine with a dose of 0.5ml/kg was determined by the age and weight of the patient.

SUMMARY:
Inguinal hernia is a common condition requiring surgical repair in the pediatric age group. The incidence of inguinal hernias is approximately 3% to 5% in term infants and 13% in infants born at less than 33 weeks of gestational age. Inguinal hernias in both term and preterm infants are commonly repaired shortly after diagnosis to avoid incarceration of the hernia. Given the lack of definitive data, optimal timing for repair of inguinal hernias in infants remains debatable[1].

: An erector spinae plane block is a relatively new regional anesthetic technique. Apart from case reports and small series, the literature regarding pediatric use is limited.

The first author to describe caudal anaesthesia as applied to children (here in connection with urologic surgical procedures) was Meredith Campbell in 1933.(2) Over time, this idea has developed into a technique of great interest, especially for use in premature infants and in newborns, considering that these paediatric subgroups are, as a result of an immature state of the CNS, at high risk of perioperative respiratory depression.

This study will be conducted to compare caudal versus ESPB as regard intraoperative and postoperative analgesia in unilateral inguinal hernia and the feasibility of ESPB in paediatric patient.

ELIGIBILITY:
Inclusion Criteria:

* age 3 moonths 6 years old
* American Society of Anesthesiologists physical status I, II for non complicated inguinal hernia.

Exclusion Criteria:

* Patients with a sepsis
* malignancy anywhere
* patient with bleeding tendencies or on anticoagulation therapy,
* allergy to study drugs
* congenital anomalies
* delayed motor or developmental milestones

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
heart rate response to skin incision | basal before surgery, after 5 minutes intra-operative, 10 minutes intra-operative, 15 minutes intra-operative
  count of heart beats per minute

SECONDARY OUTCOMES:
pain scores | at recovery, 30 minutes postoperative, 1 hour postoperative, 3 hours postoperative, 6 hours postoperative
  FLACC score at recovery FLACC score at recovery FLAAC score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicin, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided